CLINICAL TRIAL: NCT04059926
Title: National Registry of Lumen Apossing Metal Stent Incidences
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Sergio Bazaga Pérez de Rozas, Principal investigator, Hospital del Rio Hortega
Other Study IDs: RNPAL
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Interventional Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lumen metal apossing stent
  Interventions: Other: insert apossing lumen metal stent

INTERVENTIONS:
Other: insert apossing lumen metal stent — insert apossing lumen metal stent

SUMMARY:
Study design: Prospective Case Series Disease or disorder under study: Lifespan of the Axios apposition luminal prosthesis Population under study: Patients with an Axios type intraluminal apposition prosthesis

Expected dates of completion:

* Start: January 2019
* Completion: December 2020 Funding source: Does not require financing

DETAILED DESCRIPTION:
Hypothesis:

The presence of events or incidents in the follow-up and the subsequent removal of the Axios type luminal apposition prosthesis is not related to the patent time and the indication

Design:

Prospective Case Series

Methods:

- Patients: All patients who have a transmural PAL in all participating centers will be included prospectively and consecutively.

-Tracing: Patients who meet the inclusion criteria and do not present any exclusion criteria will be invited to participate in the study. The patients who agree to participate will complete the informed consent (see annex II) according to the law 41/2002 of patient autonomy without thereby altering the relationship with their doctor or causing any damage in their treatment. It will have a maximum duration of 1 year or until the first scheduled follow-up after the removal of the prosthesis. It will consist of pre-established clinical controls and radiological controls performed according to the underlying disease.

* Clinical control It will be done in person or by phone. They will be carried out after 14 days, 3, 6, 9 and 12 months from the placement of the prosthesis. Visits of 14 days, 3, 6 and 9 months may be made by telephone as an option (in case of request by the patient, limited mobility ...).
* Radiological control Radiological controls will not be performed in an established manner by participating in the study. However, abdominal imaging tests performed for any other reason will be used to confirm the presence of the stent in situ, checking these tests at the last follow-up visit.
* End of follow-up time:

A follow-up will be carried out until the first scheduled visit after the withdrawal of the PAL ( if removed at 8 weeks, it would be the 3-month visit), in patients in whom it is placed with a permanent intention, until completing 1 year of follow-up and in patients in whom technical success is not obtained until the first follow-up view (14 days). The data will be recorded in an electronic data collection notebook (CRD) in which the variables indicated in the data collection sheet will be included.

- Sample size: The number of prostheses used annually in our center ranges from 70-100. In other third level centers approximately 15-50 prostheses can be placed annually. In other centers the number of annual prostheses may be markedly lower, below the 10 annual prostheses. Depending on the number of participating centers, we consider that the number of patients included can range between 250-350.

Data management. The CRD data will be entered by the principal investigator or the collaborating researchers anonymously, encrypted and dissociated from the clinical information through a patient identification code (ID), in an online database through the RedCap platform. The responsible physician, in turn, a researcher, will define an ID for each patient, whose relationship with the medical history will only be accessible by him, with his custody in a file protected by personal password. The data entered in the database will be anonymous and the database will be password protected to which only researchers will have access.

The unified file will be kept in the Río Hortega University Hospital and will remain until the end of the study. The CRDs collected in the file will be kept in the Digestive Service to ensure their accessibility to the researchers and their control.

With regard to the application of the Organic Law on Data Protection 15/1999 and the Royal Decree 1720/2007 that develops it, it should be noted that the protocol defined in the project aimed at epidemiological analysis, determines that the files will record information completely anonymized A file will be maintained with the information collected for the development of the project within the framework defined in the Maximum Level Security Document of the Río Hortega University Hospital whose responsibility is the Management of said organization.

This document is of obligatory knowledge and available in the Intranet of the University Hospital Río Hortega. The levels of security, access and availability will be those defined in that document.

Statistical analysis. Categorical variables will be described as percentages. Continuous with normal distribution as mean and standard deviation. Continuous variables with non-normal distributions will be described as medians and interquartile range (the range can also be offered). Pearson's χ2 test or Fisher's exact test (in case the expected frequencies in the contingency tables are below 5) will be applied to assess differences between categorical variables. When analyzing possible risk factors of the objective variables (e.g., presence or absence of complications, presence or absence of embedded prostheses ...) logistic regression techniques will be used. The analysis will be carried out using Stata (StataCorp. 2013. College Station, Texas).

Ethical aspects. - Benefit-risk assessment for research subjects This study involves conducting a prospective observational study. The procedure to which patients undergo will be performed regardless of participation in the study. The only consequence of participating is that the data concerning the procedure will be collected during the procedure and that the patient will be contacted to verify the absence of deferred complications and complete the follow-up. Therefore, participation will not imply any benefit or prejudice to the participant. The benefit we hope to obtain is to identify if there are endoscopic factors that predict possible complications in the prostheses described above. This study will be carried out following the standards specified in the Declaration of Helsinki, the Standards of Good Clinical Practice, the guidelines ICH (International Conference on Harmonization) and complying with current legislation, in particular Law 14/2007 on Biomedical Research.

In cases where the placement of the prosthesis is done on a scheduled basis, prior consent will be obtained. In cases where it is performed urgently / emergently or in the face of exploration findings, consent will be requested after the exploration is completed. The principal investigator and the collaborators will be authorized to make use of the data collected in the CRD, as well as to contact the patient to complete the follow-up. In any case, the rights, security and welfare of the subjects of the study must prevail over the interests of science and society.

The patient will be identified in the study database by an identification code (ID), sex and date of birth. The databases and other documents of the study will be available to the Health Authorities if they consider it relevant, in no case will they be available to third parties.

This study will not require an insurance policy for civil liability, which covers any damages or losses derived from it.

-Data confidentiality The study data will initially be dissociated from the medical history, by means of an ID, by the responsible physician. The relationship between the ID and the medical record will be guarded by the medical researchers in a file protected with a personal password. The data will be entered in the database anonymously with the patient's ID, to maintain their anonymity. The database will be password protected, and only accessible by researchers. During the study, strict compliance with Law 15/1999, of December 13 on the Protection of Personal Data, is guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom at least the initial puncture of the access organ wall is achieved for the transmural placement of an Axios type PAL

Exclusion Criteria:

* Refusal to sign the informed consent.
* Inability to track

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have a transmural PAL are placed prospectively and consecutively
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Describe the type and proportion of complications that arise from the Axios apposition luminal prosthesis, through study completion, an average of 1 year | Through study completion, an average of 1 year
  Describe the type and proportion of complications that arise from the Axios apposition luminal prosthesis, through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vazquez-Sequeiros E, Baron TH, Perez-Miranda M, Sanchez-Yague A, Gornals J, Gonzalez-Huix F, de la Serna C, Gonzalez Martin JA, Gimeno-Garcia AZ, Marra-Lopez C, Castellot A, Alberca F, Fernandez-Urien I, Aparicio JR, Legaz ML, Sendino O, Loras C, Subtil JC, Nerin J, Perez-Carreras M, Diaz-Tasende J, Perez G, Repiso A, Vilella A, Dolz C, Alvarez A, Rodriguez S, Esteban JM, Juzgado D, Albillos A; Spanish Group for FCSEMS in Pancreas Collections. Evaluation of the short- and long-term effectiveness and safety of fully covered self-expandable metal stents for drainage of pancreatic fluid collections: results of a Spanish nationwide registry. Gastrointest Endosc. 2016 Sep;84(3):450-457.e2. doi: 10.1016/j.gie.2016.02.044. Epub 2016 Mar 10. PMID 26970012
- [Background] Siddiqui AA, Adler DG, Nieto J, Shah JN, Binmoeller KF, Kane S, Yan L, Laique SN, Kowalski T, Loren DE, Taylor LJ, Munigala S, Bhat YM. EUS-guided drainage of peripancreatic fluid collections and necrosis by using a novel lumen-apposing stent: a large retrospective, multicenter U.S. experience (with videos). Gastrointest Endosc. 2016 Apr;83(4):699-707. doi: 10.1016/j.gie.2015.10.020. Epub 2015 Oct 26. PMID 26515956
- [Background] Rinninella E, Kunda R, Dollhopf M, Sanchez-Yague A, Will U, Tarantino I, Gornals Soler J, Ullrich S, Meining A, Esteban JM, Enz T, Vanbiervliet G, Vleggaar F, Attili F, Larghi A. EUS-guided drainage of pancreatic fluid collections using a novel lumen-apposing metal stent on an electrocautery-enhanced delivery system: a large retrospective study (with video). Gastrointest Endosc. 2015 Dec;82(6):1039-46. doi: 10.1016/j.gie.2015.04.006. Epub 2015 May 23. PMID 26014960
- [Background] Kahaleh M, Shami VM, Conaway MR, Tokar J, Rockoff T, De La Rue SA, de Lange E, Bassignani M, Gay S, Adams RB, Yeaton P. Endoscopic ultrasound drainage of pancreatic pseudocyst: a prospective comparison with conventional endoscopic drainage. Endoscopy. 2006 Apr;38(4):355-9. doi: 10.1055/s-2006-925249. PMID 16680634
- [Background] Sriram PV, Kaffes AJ, Rao GV, Reddy DN. Endoscopic ultrasound-guided drainage of pancreatic pseudocysts complicated by portal hypertension or by intervening vessels. Endoscopy. 2005 Mar;37(3):231-5. doi: 10.1055/s-2005-860997. PMID 15731938
- [Background] Fabbri C, Luigiano C, Marsico M, Cennamo V. A rare adverse event resulting from the use of a lumen-apposing metal stent for drainage of a pancreatic fluid collection: "the buried stent". Gastrointest Endosc. 2015 Sep;82(3):585-7. doi: 10.1016/j.gie.2015.04.035. No abstract available. PMID 26279357
- [Background] Bang JY, Hasan M, Navaneethan U, Hawes R, Varadarajulu S. Lumen-apposing metal stents (LAMS) for pancreatic fluid collection (PFC) drainage: may not be business as usual. Gut. 2017 Dec;66(12):2054-2056. doi: 10.1136/gutjnl-2016-312812. Epub 2016 Aug 31. No abstract available. PMID 27582509
- [Background] Stecher SS, Simon P, Friesecke S, Glitsch A, Kuhn JP, Lerch MM, Mayerle J. Delayed severe bleeding complications after treatment of pancreatic fluid collections with lumen-apposing metal stents. Gut. 2017 Oct;66(10):1871-1872. doi: 10.1136/gutjnl-2016-313562. Epub 2017 Jan 12. No abstract available. PMID 28082319
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503